CLINICAL TRIAL: NCT00064909
Title: Using MR Perfusion Imaging and Hypercapnia to Study Angiogenesis in Multiple Sclerosis Patients
Brief Title: MR Perfusion Imaging and Hypercapnia (Increased Carbon Dioxide) to Study New Blood Vessel Formation in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030247; 03-CC-0247
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MRI; Perfusion; Imaging; Cerebral Blood Flow; Cerebral Blood Volume; CO2 Inhalation; Contrast Agent; Healthy Volunteer; HV
MeSH Terms: conditions — Multiple Sclerosis

SUMMARY:
This study will use magnetic resonance imaging (MRI) to examine and compare changes in blood flow and blood volume in the brains of normal volunteers and patients with multiple sclerosis (MS). Patients with MS-an inflammatory disease that attacks the brain and spine-may have new blood vessel formation (called angiogenesis) within the brain that may or may not contribute to the disease or help in repairing the brain. It is not known if these new vessels behave in the same way as the naturally occurring vessels. MRI uses a strong magnetic field and radio waves to generate brain images that provide information on brain chemistry, function, and blood flow. The results of this study may lead to a better understanding of MS.

Healthy normal volunteers and patients with multiple sclerosis 18 years of age and older may be eligible for this study. Normal volunteers must have no history of signs or symptoms of central nervous system disease. Patients with MS will be recruited from the NIH Neuroimmunology MS clinic.

All participants will undergo MRI. For this procedure, the subject lies still on a table that slides into a narrow metal cylinder (the MRI scanner). Scanning varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. During the scan, the subject wears earplugs to muffle loud knocking noises caused by electrical switching of the radio frequency circuits. The subject can communicate with the MRI staff at all times during the procedure.

During the scan, the subject wears a mask and breathes in room air or air containing 6% carbon dioxide (CO2). (Room air contains approximately 0.04% CO2, which is about 150 times less than the 6% CO2. Air that is normally breathed out contains about 5% CO2.) Breathing 6% CO2 increases the amount of blood flow in the brain that can be measured using MRI. The total duration of a single 6 percent CO2 inhalation will not exceed 10 minutes.

A catheter (thin plastic tube) is placed in a vein in the subject's arm before he or she enters the scanner. At some point during the scan, a contrast agent called gadolinium DTPA is injected into the vein through the catheter. This agent enables clearer images of the brain.

DETAILED DESCRIPTION:
Advances in MR perfusion imaging have provided clinical researchers with the opportunity to quantify regional cerebral blood flow (CBF). Recently, new vessel proliferation and formation (angiogenesis) has been observed in autopsy and biopsy specimens from patients with multiple sclerosis (MS). Newly formed MS lesions, showed strikingly increased numbers of new vessels and similar patterns were observed in and around older lesions, areas of remyelination (new myelin formation on axons, shadow plaques) and normal-appearing brain tissue. The purpose of this study is to compare CBF of MS patients, to age- and gender-matched healthy controls. CBF will be measured while subjects are inhaling room air and the increase in CBF while inhaling a mixture of room air and a known concentration of carbon dioxide (hypercapnia) will be compared. If significant new vessels growth has occurred in the brains of MS patients then this new vessel formation (neovascularization) may be reflected by a change in CBF. Comparing the CBF response to hypercapnia will determine if the newly formed vasculature includes properly functioning blood vessels. Normal cerebral blood vessels are exquisitely sensitive to the carbon dioxide in arterial blood and an increase in carbon dioxide causes CBF to increase through dilatation or relaxation of the muscles surrounding the blood vessels. In the future, changes in the hypercapnia-induced CBF response between MS patients and controls may help to monitor the treatment of the disease.

ELIGIBILITY:
INCLUSION CRITERIA (NORMAL VOLUNTEERS)

Any healthy volunteer above the age of 18 who is capable of giving informed consent recruited or self referred through the NIH Volunteer office will be eligible for this study.

All healthy normal volunteers will be required to fill out the questionnaire in Appendix B.

Normal volunteers will be included as long as they have no recorded or documented signs or symptoms of CNS disease, contraindications to an MRI and have a 'normal age-appropriate' MRI of the brain.

Only patients seen in the Neuroimmunology MS clinic with a confirmed diagnosis of Multiple Sclerosis based upon previous history of two clinical neurological attacks separated in time and in spatial location or combination of Clinical and MRI findings of a single enhancing lesion in the brain or spine along with multiple T2 hyperintensities in the juxtacortical, periventricular or infratentorial white matter according to the McDonald criteria will be included in this study.

Relapsing-remitting or secondary progressive MS who have had more than one relapse within 18 months preceding study enrollment will be recruited from the MS 7th floor clinic in the NINDS at the NIH.

MS patients EDSS score between 1.0 - 6.5, inclusive.

Give written informed consent prior to any testing under this protocol, including screening/pre-treatment tests and evaluations that are not considered part of the patient's routine care.

EXCLUSION CRITERIA:

Healthy Controls and MS patients will be excluded if they have contraindications to MR scanning, such as the following:

1. pacemakers
2. brain stimulators
3. dental implants
4. aneurysm clips (metal clips on the wall of a large artery)
5. metallic prostheses (including metal pins and rods, heart valves, and cochlear implants),
6. permanent eyeliner
7. implanted delivery pump
8. shrapnel fragments
9. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware. You will be screened for these conditions prior to the study, and if you have any of these conditions, you will not receive an MRI scan. If you have a question about any metal objects being present in your body, you should inform the physician.

Healthy controls and MS patients will be excluded from this study if they have the following:

1. History of panic disorder
2. History of migraine (because of possible complications with CO2 inhalation).
3. Subjects who have a history of a reaction to MR contrast agents specifically gadopentetate dimeglumine will be excluded from participating in the contrast agent administration part of this protocol.
4. Subjects will also be excluded from the study if they are presently taking indomethacin or acetazolamide which effects the carbonic anhydrase system of endothelial cells in the brain making them unresponsive to CO2 inhalation.
5. Subjects will be excluded if they have a previous history of panic attacks.
6. Healthy controls and MS patients will be excluded if have history of alcohol or drug abuse.
7. Healthy controls and MS patients will be excluded if concurrent, clinically significant (as determined by the investigator) cardiac, immunologic, pulmonary, neurologic, renal, and/or other major disease.
8. Healthy controls will be excluded if they have a previous known abnormality on brain MRI examination
9. Pregnant and lactating women will be excluded from the study.

MS patients will also be excluded from study entry if the following exclusion criteria exists at the time of enrollment:

1) Diagnosis of primary progressive MS, defined as gradual progression of disability from the onset without relapses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2003-07; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] van der Valk P, De Groot CJ. Staging of multiple sclerosis (MS) lesions: pathology of the time frame of MS. Neuropathol Appl Neurobiol. 2000 Feb;26(1):2-10. doi: 10.1046/j.1365-2990.2000.00217.x. PMID 10736062
- [Background] Prineas J. Pathology of the early lesion in multiple sclerosis. Hum Pathol. 1975 Sep;6(5):531-54. doi: 10.1016/s0046-8177(75)80040-2. PMID 170186